CLINICAL TRIAL: NCT03624855
Title: Implant-Associated P. Aeruginosa Bone And Joint Infections : Experience In A Regional Reference Center In France
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Research Assistant, Hospices Civils de Lyon
Other Study IDs: 18-176
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Bone and Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Description of BJI due to Pseudomonas aeruginosa: patients having bone and joint infection on implant due to Pseudomonas aeruginosa
  Interventions: Other: Bone or joint infection due to Pseudomonas aeruginosa

INTERVENTIONS:
Other: Bone or joint infection due to Pseudomonas aeruginosa — Description of bone or joint infection on implant due to Pseudomonas aeruginosa

SUMMARY:
The aim of this study is to describe the bone or joint infection due to Pseudomonas aeruginosa in patients having implant.

ELIGIBILITY:
Inclusion Criteria:

* patients having BJI on implant caused by Pseudomonas aeruginosa

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having BJI on implant caused by Pseudomonas aeruginosa managed at the Croix Rousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Description and rate of bone or joint infection on implant caused due to Pseudomonas aeruginosa | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Description of the type of infection due to P. aeruginosa : patients and type of implant, profile of the bacterium, medical and chirurgical treatment, rate

SECONDARY OUTCOMES:
Rate of adverse events occurring under medical treatment against Pseudomonas aeruginosa | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  description of adverse events occurring under medical treatment against Pseudomonas aeruginosa in BJI
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, Md,PhD, Principal Investigator — Hospices Civils de Lyon Hôpital de la Croix-Rousse
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided